CLINICAL TRIAL: NCT01252719
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Single-Dose IV Oritavancin Versus IV Vancomycin for the Treatment of Patients With Acute Bacterial Skin and Skin Structure Infection (SOLO I)
Brief Title: Oritavancin Versus IV Vancomycin for the Treatment of Participants With Acute Bacterial Skin and Skin Structure Infection (SOLO I)
Acronym: SOLO I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMC-ORI-10-01
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Wound Infection; Abscess; Systemic Inflammation; Cellulitis
Keywords: ABSSSI; Skin Infection; Abscess
MeSH Terms: conditions — Wound Infection; Abscess; Cellulitis | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-Dose IV Oritavancin Diphosphate (Experimental)
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate; Drug: Placebo
- IV Vancomycin (Active Comparator)
  Interventions: Drug: IV Vancomycin

INTERVENTIONS:
Drug: Single-Dose IV Oritavancin Diphosphate — Oritavancin was administered as a single IV dose.
  Arms: Single-Dose IV Oritavancin Diphosphate
Drug: IV Vancomycin — Intravenous vancomycin was administered for a minimum of 7 days and up to a maximum of 10 days.
  Arms: IV Vancomycin
Drug: Placebo — Intravenous placebo was administered thereafter, for a minimum of 7 days and up to a maximum of 10 days (oritavancin and placebo).
  Arms: Single-Dose IV Oritavancin Diphosphate

SUMMARY:
The purpose of this Phase 3 trial was to evaluate the efficacy, safety, and tolerability of oritavancin in acute bacterial skin and skin structure infections (ABSSSIs), including those caused by methicillin-resistant staphylococcus aureus (MRSA), and to evaluate the potential economic benefit of oritavancin administered as a single 1200-milligram (mg) intravenous (IV) dose.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, parallel, comparative efficacy and safety study of single-dose IV oritavancin/IV placebo versus IV vancomycin for 7 to 10 days in adults with ABSSSI suspected or proven to be caused by gram-positive pathogens. Approximately 960 participants were to be randomized at 100 centers globally.

In addition, this study characterized the pharmacokinetics (PK) and PK/pharmacodynamics (PD) properties of a single 1200-mg IV dose of oritavancin and evaluated the potential health economic benefits offered by this dosing strategy.

ELIGIBILITY:
Inclusion Criteria:

Participants were included in the study if they met all of the following inclusion criteria:

1. Males or females ≥18 years old
2. Diagnosis of ABSSSI suspected or confirmed to be caused by a gram-positive pathogen requiring at least 7 days of IV therapy
3. An ABSSSI included 1 of the following infections: wound infections, cellulitis/erysipelas, major cutaneous abscess
4. ABSSSI must have presented with at least 2 local signs and symptoms and at least 1 sign of systemic inflammation (unless >70 years of age).
5. Able to give informed consent and willing to comply with all required study procedures

Exclusion Criteria:

Participants were excluded from the study if any of the following exclusion criteria applied prior to randomization:

1. Prior systemic or topical antibacterial therapy with activity against suspected or proven gram-positive pathogens within the preceding 14 days unless:

   * The causative gram-positive pathogen(s) isolated from the ABSSSI site was/were resistant in vitro to the antibacterial(s) that was/were administered with documented clinical progression.
   * Documented failure to previous ABSSSI antibiotic therapy was available. Documentation of treatment failure must have been recorded.
   * Participant received a single dose of a short-acting antibacterial therapy 3 or more days before randomization.
2. Infections associated with, or in close proximity to, a prosthetic device
3. Severe sepsis or refractory shock
4. Known or suspected bacteremia at time of Screening
5. ABSSSI due to or associated with any of the following:

   * Infections suspected or documented to be caused by gram-negative pathogens
   * Wound infections (surgical or traumatic) and abscesses with only gram-negative pathogens
   * Diabetic foot infections
   * Concomitant infection at another site not including a secondary ABSSSI lesion
   * Infected burns
   * A primary infection secondary to a pre-existing skin disease with associated inflammatory changes
   * Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease
   * Any evolving necrotizing process gangrene or infection suspected or proven to be caused by Clostridium species
   * Infections known to be caused by a gram-positive organism with a vancomycin minimum inhibitory concentration >2 micrograms/milliliter or clinically failing prior therapy with glycopeptides
   * Catheter site infections
6. Allergy or intolerance to aztreonam or metronidazole in a participant with suspected or proven polymicrobial wound infection involving gram-negative and/or anaerobic bacteria
7. Was currently receiving chronic systemic immunosuppressive therapy
8. Acquired immunodeficiency syndrome with cluster of differentiation 4 count <200 cells/cubic millimeter
9. Neutropenia
10. Significant or life-threatening condition that would confound or interfere with the assessment of the ABSSSI
11. Women who were pregnant or nursing
12. History of immune-related hypersensitivity reaction to glycopeptides
13. Participants that required anticoagulant monitoring with an activated partial thromboplastin time
14. Contraindication to vancomycin
15. Participants unwilling to forego blood and/or blood product donation
16. Treatment with investigational medicinal product within 30 days before enrollment and for the duration of the study
17. Investigational device present, or removed <30 days before enrollment, or presence of device-related infection
18. Participants unlikely to adhere to the protocol, comply with study drug administration, or complete the clinical study
19. Severe hepatic disease
20. Presence of hyperuricemia
21. Unwilling to refrain from chronic use of any medication with antipyretic properties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Sharp Chula Vista Medical Center, Chula Vista, California, United States

REFERENCES:
- [Derived] Corey GR, Loutit J, Moeck G, Wikler M, Dudley MN, O'Riordan W; SOLO I and SOLO II investigators. Single Intravenous Dose of Oritavancin for Treatment of Acute Skin and Skin Structure Infections Caused by Gram-Positive Bacteria: Summary of Safety Analysis from the Phase 3 SOLO Studies. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e01919-17. doi: 10.1128/AAC.01919-17. Print 2018 Apr. PMID 29358292
- [Derived] Deck DH, Jordan JM, Holland TL, Fan W, Wikler MA, Sulham KA, Ralph Corey G. Single-Dose Oritavancin Treatment of Acute Bacterial Skin and Skin Structure Infections: SOLO Trial Efficacy by Eron Severity and Management Setting. Infect Dis Ther. 2016 Sep;5(3):353-61. doi: 10.1007/s40121-016-0119-9. Epub 2016 Jul 1. PMID 27370913
- [Derived] Corey GR, Kabler H, Mehra P, Gupta S, Overcash JS, Porwal A, Giordano P, Lucasti C, Perez A, Good S, Jiang H, Moeck G, O'Riordan W; SOLO I Investigators. Single-dose oritavancin in the treatment of acute bacterial skin infections. N Engl J Med. 2014 Jun 5;370(23):2180-90. doi: 10.1056/NEJMoa1310422. PMID 24897083

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-Dose 1200 mg Oritavancin: Single 1200 milligram (mg) intravenous (IV) dose of oritavancin diphosphate administered as first infusion followed by IV placebo administered twice daily for a minimum of 7 days and up to a maximum of 10 days.
- Vancomycin: Intravenous vancomycin, 1 gram (g) or 15 mg/kilogram (kg), administered twice daily for a minimum of 7 days and up to a maximum of 10 days.
Period: Overall Study
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Started | 483 (Participants Randomized) | 485 (Participants Randomized)
Modified Intent to Treat Population | 475 | 479
Completed | 433 | 423
Not Completed | 50 | 62

BASELINE CHARACTERISTICS:
Population: Modified intent to treat (mITT) population consisting of all participants who were randomized into the trial and received any study drug.
Groups:
- Single-Dose 1200 mg Oritavancin: Single 1200 mg IV dose of oritavancin diphosphate administered as first infusion followed by IV placebo administered twice daily for a minimum of 7 days and up to a maximum of 10 days.
- Vancomycin: Intravenous vancomycin, 1 g or 15 mg/kg, administered twice daily for a minimum of 7 days and up to a maximum of 10 days.
- Total: Total of all reporting groups
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin | Total
Number analyzed (Participants) | 475 | 479 | 954
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.20) | 44.3 (14.50) | 45.2 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 178 | 352
  Male | 301 | 301 | 602

OUTCOME MEASURES:

1. Secondary Outcome: Investigator Assessed Clinical Cure Of Treatment With Single-dose IV Oritavancin Compared With IV Vancomycin For 7 To 10 Days At Post-therapy Evaluation (Key Secondary Endpoint)
Description: Compared the clinical efficacy at the post therapy evaluation of oritavancin and vancomycin based on the Investigator examination of the signs and symptoms of the primary acute bacterial skin and skin structure infection (ABSSSI). Investigator assessment of clinical cure was complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics was needed.
Time Frame: 7-14 days after end of therapy
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 475 | 479
participants
  Clinical Cure | 378 | 383
  Clinical Failure | 97 | 96
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test was a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the two-sided 95% CI for the difference in response rates in the mITT population was greater than -10%, the NI of oritavancin to vancomycin was concluded; Difference in Proportions = -0.4, 95% CI 2-sided [-5.5 to 4.7]

2. Primary Outcome: Cessation Of Spread Or Reduction In Size Of Baseline Lesion, Absence Of Fever, And No Rescue Antibiotic Medication At Early Clinical Evaluation (ECE) (48 To 72 Hours)
Description: Clinical response at the ECE visit (48-72 hours following initiation of study drug administration). Early clinical response was defined as a composite outcome based on cessation of spreading or reduction in the size of baseline lesion, absence of fever and no rescue antibiotic medication.
  A participant was classified as "success" if all of the following were met: cessation of spread or reduction of the lesion (defined as cessation of spread of the redness, edema, and/or induration or reduction in size [length, width, and area] of the redness, edema, and/or induration such that the size of the lesion was less than or equal to the size at baseline); resolution (absence) of fever (temperature <37.7°Celsius at the last 3 consecutive recordings by the same route of administration taken 4 times per day, for example every 6 hours between 48 and 72 hours); no rescue antibiotic medication.
Time Frame: 48-72 hours after the initiation of study therapy
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 475 | 479
participants
  Success | 391 | 378
  Failure | 84 | 101
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test was a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the two-sided 95% confidence interval (CI) for the difference in response rates in the mITT population was greater than -10% the non-inferiority (NI) of oritavancin to vancomycin was concluded; Difference in Proportions = 3.4, 95% CI 2-sided [-1.6 to 8.4]

3. Secondary Outcome: Number Of Participants With A Lesion Size Reduction ≥20% From Baseline At ECE
Description: Clinical response at the ECE visit (48-72 hours following initiation of study drug administration) based on changes in ABSSSI lesion size measurements from baseline. Participants with a ≥20% reduction in size of baseline lesion were classified a 'success', while those with missing data or those without a reduction in size of baseline lesion ≥20% were classified a 'failure'.
Time Frame: 48-72 hours after the initiation of study therapy
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 475 | 479
Participants
  Success | 413 | 397
  Failure | 62 | 82
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test was a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the two-sided 95% CI for the difference in response rates in the mITT population was greater than -10% the NI of oritavancin to vancomycin was concluded; Difference in Proportions = 4.1, 95% CI 2-sided [-0.5 to 8.6]

ADVERSE EVENTS:
Time Frame: Begins from the time the participant provided informed consent through to the last follow-up visit at 60 (+7) days.
Description: Adverse events were analyzed in the safety population consisting of all participants who received any study drug. The analysis was performed according to the actual treatment that the participant received.
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
All-Cause Mortality (participants affected / at risk) | 1/473 | 2/481
Serious Adverse Events (participants affected / at risk) | 35/473 | 35/481
Other Adverse Events (participants affected / at risk) | 323/473 | 340/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Dose 1200 mg Oritavancin (N=473) | Vancomycin (N=481)
Cellulitis (Infections and infestations) | 5 | 8
Skin Infection (Infections and infestations) | 3 | 1
Subcutaneous abscess (Infections and infestations) | 3 | 1
Abscess limb (Infections and infestations) | 3 | 0
Abscess (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Skin bacterial infection (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Periorbital access (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Serum sickness-like reaction (Immune system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Infusion site thrombosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Dose 1200 mg Oritavancin (N=473) | Vancomycin (N=481)
Nausea (Gastrointestinal disorders) | 52 | 43
Vomiting (Gastrointestinal disorders) | 23 | 18
Headache (Nervous system disorders) | 34 | 38
Diarrhea (Gastrointestinal disorders) | 23 | 17
Cellulitis (Infections and infestations) | 20 | 17
Infusion site reaction (General disorders) | 19 | 34
Constipation (Gastrointestinal disorders) | 19 | 21
Infusion site extravasation (General disorders) | 18 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 44
Pyrexia (General disorders) | 15 | 20
Dizziness (Nervous system disorders) | 15 | 15
Insomnia (Psychiatric disorders) | 14 | 13
Abscess limb (Infections and infestations) | 13 | 5
Pruritus generalized (Skin and subcutaneous tissue disorders) | 11 | 9
Alanine aminotransferase increased (Investigations) | 11 | 5
Chills (General disorders) | 10 | 12
Fatigue (General disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and PI agree that the Sponsor shall have the right to the first publication of the Study results. The Pl may publish data or results from the Study; provided, however, that the Institution and/or PI submits the proposed publication to Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary.